CLINICAL TRIAL: NCT05235087
Title: Bovine Atelocollagen Skin Sensitization Test
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: AscentX Medical's business strategy changed.
Sponsor: AscentX Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 21-ASMI-101
Record Dates: First submitted 2022-01-27; First posted 2022-02-10 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Bovine Atelocollagen Skin Sensitization Test (Experimental): Volunteer cohort tested for hypersensitivity towards intradermal injection of bovine atelocollagen.
  Interventions: Device: Bovine atelocollagen intradermal injection

INTERVENTIONS:
Device: Bovine atelocollagen intradermal injection — Intradermal skin test injection

SUMMARY:
Bovine atelocollagen skin testing of healthy adult volunteers to investigate the potential of allergy to atelocollagen medical device implants

DETAILED DESCRIPTION:
Day 01: Receive 0.1 mL intradermal injection of atelocollagen skin test into left volar forearm.

Day 15: Receive 2nd intradermal injection of 0.1 mL atelocollagen skin test into right volar forearm (14 days after 1st injection).

Day 45: Final assessment of both injection sites (30 days after 2nd injection)

Note: ALL injection sites will be assessed clinically at 30 minutes (for observational purposes) and at 72 hours (to determine response) after each injection. Visit windows for 72 hour assessments, and Day 15 and Day 45 visits can occur up to 96 hours (4 days) after target time.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers, of either sex, aged at least 18 years.
* Volunteers must be capable of understanding and following directions in English.
* Subjects who are healthy and have normal skin on the volar surface of the forearm.
* Subjects willing and able to comply with the requirements of the study.
* Subjects willing and able to comply with the follow-up requirements.
* Subjects willing and able to give written and verbal informed consent.

Exclusion Criteria:

* Subjects who are pregnant, nursing or intend to become pregnant.
* Current treatment by a physician for allergy, unless physician consulted by Investigator and participation was approved.
* Participation in a repeat insult patch test (RIPT), skin prick test (SPT) or follow-up work within the last month.
* Recent immunization, including COVID-19 (less than 14 days prior to skin test).
* Subjects who have had any form of collagen soft tissue treatment within the last 12 months.
* Subjects with medical history indicating atopy or dermatographia ('skin writing').
* Subject has a current skin disease of any type apart from mild facial acne (e.g., eczema, psoriasis).
* Subject has any skin pathology or condition that could interfere with the evaluation of the treatment areas.
* Subjects who were or are currently being treated with any systemic immuno-suppressive therapy, including but not limited to chemotherapy agents or cortico-steroids (including inhaled or insufflated) within the past 3 months.
* Subjects who were or are currently being treated with any topical OTC drug or prescription therapy on their arms (below the elbow) within the past 3 months.
* Subjects with a history indicative of abnormal immune function (e.g., auto- immune diseases, HIV, cancer, etc.).
* Subjects with known lidocaine hypersensitivity.
* Subjects with known sensitivity to bovine collagen.
* Subjects who have a history of dietary beef allergy, undergoing desensitization to beef products or planning to undergo desensitization within the study evaluation period.
* Subjects with severe allergies manifested by a history of anaphylaxis.
* Subject is currently enrolled in an investigational drug or device study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2023-11-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Hypersensitivity Evaluation | 44 days
  Subjects will monitor the implant sites daily for signs of local reactions and are instructed to record other clinical symptoms occurring during the course of the study. Unscheduled visits will be secured if subjects report adverse events between scheduled visits. Hypersensitivity to the xenogenic collagen test material will be assessed through visual scoring by trained clinical staff, a qualified physician, and subject diary observations. All potential reactions will be photographed by study staff for scoring confirmation.
  Hypersensitivity reaction will be assessed based on FDA's recent draft guidance "Assessing the Irritation and Sensitization Potential of Transdermal and Topical Delivery Systems for ANDAs. A positive response is defined as a skin response greater than Score 2 of 4 mm diameter at the implant site persisting more than 72 hours, with photograph, and verification of an immune reaction by histopathology of the site biopsy.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Rullan, MD, Principal Investigator — Dermatology Institute
Locations (1):
- Dermatology Institute, Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cooperman LS, Mackinnon V, Bechler G, Pharriss BB. Injectable collagen: a six-year clinical investigation. Aesthetic Plast Surg. 1985;9(2):145-51. doi: 10.1007/BF01570347. PMID 3161303
- [Background] Lynn AK, Yannas IV, Bonfield W. Antigenicity and immunogenicity of collagen. J Biomed Mater Res B Appl Biomater. 2004 Nov 15;71(2):343-54. doi: 10.1002/jbm.b.30096. PMID 15386396
- [Background] Velosa APP, Brito L, de Jesus Queiroz ZA, Carrasco S, Tomaz de Miranda J, Farhat C, Goldenstein-Schainberg C, Parra ER, de Andrade DCO, Silva PL, Capelozzi VL, Teodoro WR. Identification of Autoimmunity to Peptides of Collagen V alpha1 Chain as Newly Biomarkers of Early Stage of Systemic Sclerosis. Front Immunol. 2021 Feb 12;11:604602. doi: 10.3389/fimmu.2020.604602. eCollection 2020. PMID 33643291
- [Background] Pendaries V, Gasc G, Titeux M, Leroux C, Vitezica ZG, Mejia JE, Decha A, Loiseau P, Bodemer C, Prost-Squarcioni C, Hovnanian A. Immune reactivity to type VII collagen: implications for gene therapy of recessive dystrophic epidermolysis bullosa. Gene Ther. 2010 Jul;17(7):930-7. doi: 10.1038/gt.2010.36. Epub 2010 Apr 8. PMID 20376098
- [Background] Ujiie H, Yoshimoto N, Natsuga K, Muramatsu K, Iwata H, Nishie W, Shimizu H. Immune Reaction to Type XVII Collagen Induces Intramolecular and Intermolecular Epitope Spreading in Experimental Bullous Pemphigoid Models. Front Immunol. 2019 Jun 19;10:1410. doi: 10.3389/fimmu.2019.01410. eCollection 2019. PMID 31275329
- [Background] Daniels, et al. Process for augmenting connective mammalian tissue with in situ polymerizable native collagen solution. US 3,949,073, United States Patent and Trademark Office, 6 April 1976.
- [Background] Luck, et al. Aqueous collagen composition. US 4,140,537, United States Patent and Trademark Office, 20 February 1979.
- [Background] Luck, et al. Non-antigenic collagen and articles of manufacture. US 4,233,360, United States Patent and Trademark Office, 11 November 1980.
- [Background] Smestad, et al. Injectable cross-linked collagen implant material. US 4,582,640, United States Patent and Trademark Office, 15 April 1986
- [Background] Cohen S, Dover J, Monheit G, Narins R, Sadick N, Werschler WP, Karnik J, Smith SR. Five-Year Safety and Satisfaction Study of PMMA-Collagen in the Correction of Nasolabial Folds. Dermatol Surg. 2015 Dec;41 Suppl 1:S302-13. doi: 10.1097/DSS.0000000000000542. PMID 26618457
- [Background] Cohen SR, Holmes RE. Artecoll: a long-lasting injectable wrinkle filler material: Report of a controlled, randomized, multicenter clinical trial of 251 subjects. Plast Reconstr Surg. 2004 Sep 15;114(4):964-76; discussion 977-9. doi: 10.1097/01.prs.0000133169.16467.5f. PMID 15468406
- See also: Zyderm® highly purified dermal collagen implant — https://www.rxlist.com/zyderm-drug.htm#description
- See also: BellaFill® Skin Test Instructions for Use (PN: 7252 Rev 00 (10/2018)) — http://www.bellafill.com
- See also: ArteFill® FDA Summary of Safety and Effectiveness (2006) — https://www.accessdata.fda.gov/cdrh_docs/pdf2/P020012b.pdf